CLINICAL TRIAL: NCT05441930
Title: An Interventional, Open Label, Controlled, Randomized, Pairwise, Phase Ib Safety, Tolerability and Pharmacokinetic (PK) Study of Levofloxacin Ocular Implant in Patients Undergoing Routine Bilateral Cataract Surgery
Brief Title: A Study of Levofloxacin Ocular Implant in Patients Undergoing Routine Bilateral Cataract Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor has suspended study to conserve capital for clinical development of lead asset
Sponsor: PolyActiva Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVO-CS102
Record Dates: First submitted 2022-06-19; First posted 2022-07-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Once eligible, subject eyes will be randomized to determine which eye will receive the first surgery. After the first surgery, study participants will receive the control treatment consisting of commercially available topical medications. For the second cataract surgery, study participants will receive a single Levofloxacin Ocular Implant in the posterior sulcus in the surgical eye at the end of cataract surgery. No sham dosing will be conducted in the eyes in the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levofloxacin Ocular Implant (Experimental): Biphasic levofloxacin antibiotic implant
  Interventions: Drug: Levofloxacin Ocular Implant
- Control (Active Comparator): Commercially available topical medications as per LEVO-CS102 Surgical Therapy Procedure.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Levofloxacin Ocular Implant — Levofloxacin Ocular Implant an implant that delivers a bolus dose of levofloxacin and a constant daily dose for a further 5-7 days.
  Arms: Levofloxacin Ocular Implant
Drug: Control — Commercially available topical medications as per LEVO-CS102 Surgical Therapy Procedure.
  Arms: Control

SUMMARY:
Open label controlled interventional study in eyes in up to 12 subjects (24 eyes) scheduled for uncomplicated bilateral cataract surgery on separate days.

DETAILED DESCRIPTION:
This is a multicenter, open label, controlled, pairwise, interventional study in eyes in up to 12 subjects (24 eyes) scheduled for uncomplicated bilateral cataract surgery on separate days. Eligible individuals provide informed consent; and are screened for inclusion in the study.

Once eligible, subject eyes will be randomized to determine which eye will receive the first surgery. After the first surgery, study participants will receive the control treatment consisting of commercially available topical medications. For the second cataract surgery, study participants will receive a single Levofloxacin Ocular Implant in the posterior sulcus in the surgical eye at the end of cataract surgery. No sham dosing will be conducted in the eyes in the control arm.

ELIGIBILITY:
Key Inclusion Criteria

1. Male or female subjects 18 years of age or older.
2. Willing and able to understand and sign an informed consent form prior to any study-related procedures.
3. Willing and able to follow study instructions, and able to be present for the required study visits/assessments for the duration of the study.
4. Diagnosis of cataract in both eyes scheduled for sequential bilateral elective cataract extraction by phacoemulsification and posterior chamber IOL implantation not combined with any other surgery except femtosecond laser.
5. Minimum endothelial cell density (ECD) in both eyes of greater than or equal to 2000 cells per mm2.
6. Fully vaccinated against COVID-19, as evidenced by vaccination record.

Key Opthalmic Exclusion Criteria

Ophthalmic:

1. Have a history of or current uveitis, macular edema (cystoid or diabetic), diabetic retinopathy, retinal vein occlusion and neovascular glaucoma, corneal conditions such as keratitis, corneal edema or advanced macular degeneration, which in the opinion of the investigator would interfere with study assessments and confound the data.
2. In the opinion of the investigator or reading center, have confluent central corneal guttatae, multiple central guttatae greater than a single cell, or corneal disease or abnormality that would prevent specular microscopy corneal scans.
3. Aphakia or low vision or monocular.
4. Have had any intraocular surgery, glaucoma surgery (including but not limited to filtering surgery like trabeculectomy, Ahmed valve, etc) or cornea/refractive surgery within the past 6 months or anticipate a need for eye surgery (including laser) during the study period.
5. Use of prostaglandin (PG) analogues within 60 days prior to Screening or during the course of the study.
6. Subjects with clinically diagnosed Fuchs' Endothelial Corneal Dystrophy (FECD)/ history of keratoplasty.
7. Subjects for whom an intra-ocular or glaucoma device procedure is planned during the cataract procedure, during study participation or has been previously undertaken.
8. Have a current retinal detachment or history of blunt trauma in either eye.
9. Subject who in the opinion of the surgeon has a high risk of the posterior capsule being compromised/zonular dehiscence during cataract surgery.
10. Intraoperative complications during the cataract surgery including posterior capsule rupture, zonular dehiscence, non-placement of Posterior Chamber Intra Ocular Lens (PCIOL), vitreous prolapse, lens fragments in the vitreous, placement of Anterior Chamber Intra Ocular Lens (ACIOL), uncontrolled bleeding /hyphema.
11. Known sensitivity to any component of the product (e.g. fluoroquinolone or polyurethane sensitivity), or to topical therapy used during course of study (e.g., povidone iodine, or anesthetics).
12. Used fluoroquinolone antibiotics (topically, orally or systemically) during the 4 weeks before screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-23 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-14 (Estimated)

PRIMARY OUTCOMES:
Safety of the Levofloxacin Ocular Implant | Day 90
  Descriptive summary statistics will be used to assess the number and frequency of ocular and non ocular adverse events
Levofloxacin concentration in aqueous humor at Day 5 in treated eyes | Day 5
  To determine levofloxacin concentration in aqueous humor at Day 5 in eyes with the Levofloxacin Ocular Implant to facilitate dose adjustment for Phase II studies.

SECONDARY OUTCOMES:
Number of actuations required to administer the implant | Day 0
  Clinicians administering the implant will record the number of actuations required to use the custom-built administration device

CONTACTS AND LOCATIONS:
Overall Officials: Michael Coote, MD, Principal Investigator — Melbourne Eye Specialists
Locations (3):
- United States (2):
  - Ophthalmology Associates, St Louis, Missouri
  - Carolina Cataract and Laser Centre, Ladson, South Carolina
- Melbourne Eye Specialists, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No